CLINICAL TRIAL: NCT04782687
Title: A Phase II Trial of Daratumumab, Lenalidomide and Dexamethasone (DRd) in Combination With Selinexor for Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Study of Selinexor Plus DRd for Newly Diagnosed Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20285; IST-337 (Other: Karyopharm Therapeutics, Inc)
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma; Myeloma Multiple; Kahler Disease; Myeloma, Plasma Cell; Myeloma-Multiple; Myelomatosis; Plasma Cell Myeloma
Keywords: myeloma; cancer; newly diagnosed multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Neoplasms | interventions — selinexor; Dexamethasone; daratumumab; Lenalidomide

STUDY DESIGN:
Intervention Model Description: This is a single-arm, phase II, open-label, non-blinded, trial to investigate the effects of S-DRd for first line treatment of multiple myeloma in patients who are ineligible for stem cell transplant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Selinexor plus DRd (Experimental): 1. Lenalidomide 15 mg orally on Days 1-21 of each 28-day cycle
  2. Dexamethasone 40 mg on Days 1, 8, 15, 22 of each cycle. However, those >75 years old may be administered a weekly dose of 20 mg dexamethasone.
  3. Daratumumab 1800 mg subcutaneous injection once weekly in Cycles 1 and 2, every 2 weeks in cycles 3 to 6, and every 4 weeks thereafter.
  4. Selinexor 60 mg on Days 1, 8, 15, of cycles 1-3, with a planned dose-reduction to 40 mg on Days 1, 8, 15 for cycles beyond 3. If patient was previously dose reduced prior to cycle 4, then at cycle 4 planned dose reduction, you will again decrease dose by 1 level.
  Interventions: Drug: Selinexor; Drug: Dexamethasone Oral; Drug: Daratumumab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Selinexor — oral drug that comes in 20 mg tablets
  Other Names: Xpovio
Drug: Dexamethasone Oral — Dexamethasone 40 mg on Days 1, 8, 15, 22 of each cycle. However, those >75 years old may be administered a weekly dose of 20 mg dexamethasone.
Drug: Daratumumab — Patients will receive daratumumab subcutaneously (SC, or under the skin) as an injection. The recommended dosage of the SC formulation is 1,800 mg daratumumab and 30,000 units hyaluronidase administered SC into the abdomen over approximately 3 to 5 minutes according to recommended schedule.
  Daratumumab 1800 mg subcutaneously once weekly in Cycles 1 and 2, every 2 weeks in cycles 3 to 6, and every 4 weeks thereafter.
  Other Names: Darzalex
Drug: Lenalidomide — Patients will receive a 21-day supply of lenalidomide (15 mg) as oral capsules, as appropriate, for each 28-day treatment cycle
  Other Names: Revlimid

SUMMARY:
This is a single-arm, phase II, open-label trial to investigate the effects of selinexor (S) in combination with daratumumab, lenalidomide, and dexamethasone (DRd) for first-line treatment of multiple myeloma (MM).

FDA has approved selinexor plus dexamethasone in multiple myeloma after four prior therapies, and DRd is also already approved by the FDA for multiple myeloma. This study will use all four (S-DRd) together to treat MM as an initial treatment.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is an incurable disease with high death rates as a result of developing resistance to treatments. Even with the advent of novel therapies, myeloma patients ultimately progress from frontline therapy. Common treatments include glucocorticoids, chemotherapy, proteasome inhibitors (PIs), Immunomodulatory imide drugs (IMiDs), stem cell transplants, and radiation therapy. Optimal frontline therapy with deeper remissions translates to improved overall survival and progression free survival. The purpose of this study is to investigate and improve upon reported outcomes in the frontline setting.

Selinexor has shown potent anti-myeloma activity in preclinical models of MM and Phase 1, Phase 2 clinical studies as well as in a randomized phase 3 clinical trial called BOSTON. Selinexor was approved by the US FDA in July 2019 in combination with dexamethasone for the treatment of adult patients relapsed/refractory (RR) MM who have received at least four prior therapies and whose disease is refractory to at least two proteasome inhibitors, at least two immunomodulatory agents, and an anti-CD38 (anti-cluster of differentiation 38) monoclonal antibody. In June 2020, Selinexor was approved as a monotherapy by the FDA for adult patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) after at least 2 lines of systemic therapy.

Treatment with combination therapies including daratumumab, lenalidomide, and dexamethasone has shown improvement in response rates, time to progression, and survival. Daratumumab is an approved CD38-directed cytolytic antibody used as a monotherapy for patients with heavily pre-treated MM, and in combination with lenalidomide and dexamethasone. The risk of death or disease progression was 44% lower and increased overall response rate (ORR) of 92.9% was observed in patients with newly diagnosed MM that received the triplet combination of daratumumab, lenalidomide, and dexamethasone (DRd) compared to lenalidomide and dexamethasone alone (Rd).

Tolerability of the DRd combination in patients was consistent between DRd and Rd treatments. The safety profile of DRd was shown to be consistent with known safety profiles of daratumumab and Rd. Higher rates of infections (upper respiratory tract infection and pneumonia) and neutropenia in DRd treated patients than in Rd treated patients were observed. However, grade 3 or 4 infections were similar between DRd and Rd treatment groups and were managed by standard of care. After exposure to DRd for a median of 34 months, no new safety concerns were observed in the extended follow-up of the POLLUX phase III study.

Preclinical data demonstrated that patient-derived MM cells were sensitized to the combination of Selinexor and daratumumab compared to the single agents. Clinical data demonstrate an ORR of 74% in patients with relapsed myeloma treated with Selinexor, daratumumab, and dexamethasone.

The rationale for the combination of Selinexor, lenalidomide, daratumumab, and dexamethasone (S-DRd) in the current study is based on the following: preclinical synergistic activities observed with Selinexor and dexamethasone, the preclinical activity of Selinexor combined with both lenalidomide and daratumumab; as well as the clinical experience of the combination of Selinexor and lenalidomide/dexamethasone can be safely combined with 92% ORR in patients with relapsed myeloma; and the combination of Selinexor and daratumumab/dexamethasone can also be safely combined with an ORR of 74%. There is an urgent need to induce more efficient, deeper and durable responses in patients with newly diagnosed MM.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Have documented multiple myeloma as defined by the International Myeloma Working Group (IMWG) 2015 criteria below:

   Clonal bone marrow plasma cells ≥10% or biopsy-proven bony or extramedullary plasmacytoma. * In addition, the patient must meet one of the criteria in either 2a or 2b.
   1. Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically at least one of the following:

      * i. Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than the upper limit of normal (ULN) or >2.75 mmol/L (>11 mg/dL)
      * ii. Renal insufficiency: creatinine clearance 20-40 mL per min or serum creatinine >177 μmol/L (>2 mg/dL)
      * iii. Anemia: hemoglobin value of > 2 g/dL below the lower limit of normal, or a hemoglobin value <10 g/dL*
      * iv. Bone lesions: one or more osteolytic lesions on skeletal radiography, or CT (computed tomography) **.
   2. Any one or more of the following:

      * i. Clonal bone marrow plasma cell percentage* ≥60%
      * ii. Involved: uninvolved serum free light chains (FLC) ratio*** >100
      * iii. >1 focal lesions on MRI (magnetic resonance imaging) studies; Each focal lesion must be 5 mm or more in size.
      * Clonality should be established by showing κ/λ-light-chain restriction on flow cytometry, immunohistochemistry, or immunofluorescence. Bone marrow plasma cell percentage should preferably be estimated from a core biopsy specimen; in case of a disparity between the aspirate and core biopsy, the highest value should be used.
      * If bone marrow has less than 10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement.
      * These values are based on the serum Freelite assay. The involved FLC must be ≥100 mg/L.
3. Have measurable disease as defined by any of the following:

   1. Serum M-protein level ≥0.5 g/dL or urine M protein level ≥200 mg/24 hours; or
   2. Immunoglobulins A, D, E or M multiple myeloma: serum M-protein level ≥0.5 g/dL or urine M-protein level ≥200 mg/24 hours; or
   3. Light chain multiple myeloma without measurable disease in the urine: serum Ig FLC ≥10 mg/dL and abnormal serum Ig kappa/lambda FLC ratio
4. Have previously untreated myeloma. For previously untreated patients an emergency course of steroids (defined as no greater than 40 mg of dexamethasone, or equivalent per day for a maximum of 4 days) is permitted. In addition, radiation therapy is permitted prior to study entry, during screening, and during study treatment as needed for lytic bone disease.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
6. Female patients of childbearing potential must have a negative serum pregnancy test at screening and agree to use highly effective methods of contraception throughout the study and for 90 days following the last dose of study treatment. Childbearing potential excludes: Age >50 years and naturally amenorrhoeic for >1 year, or previous bilateral salpingo-oophorectomy, or hysterectomy.
7. Male patients who are sexually active must use highly effective methods of contraception throughout the study and for 3 months after receiving the last dose of study drug. Male patients must agree not to donate sperm during the study treatment period and for 3 months after receiving the last dose of study drug.
8. Patients must be willing and able to adhere to the prohibitions and restrictions specified in this protocol and referenced in the informed consent form (ICF).
9. Each patient (or their legally acceptable representative) must sign an ICF indicating that he or she understands the purpose of, and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. Exhibiting clinical signs of or has a known history of meningeal or central nervous system involvement by multiple myeloma.
2. Is known to be seropositive for human immunodeficiency virus, known to have hepatitis B surface antigen positivity, or known to have a history of hepatitis C.

   Patients who completed treatment for hepatitis C and have no detectable circulating hepatitis C virus (HCV) by hepatitis C RNA polymerase chain reaction (PCR) for at least 6 months prior to screening, may participate in the study. Such patients will be required to undergo regular assessment for HCV reactivation during their participation in the study. Patients who test positive for HCV at any time during these assessments will be withdrawn from the study.
3. Has any concurrent medical condition or disease (e.g., active systemic infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.
4. Has clinically significant cardiac disease, including:

   * Myocardial infarction (MI) within 6 months before first day of first cycle (C1D1), or unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV)
   * Uncontrolled cardiac arrhythmia (NCI-CTCAE Version 5.0 Grade 2 or higher) or clinically significant electrocardiogram (ECG) abnormalities
5. Screening 12-lead ECG shows a baseline QT interval (QTc) >470 msec
6. Has any of the following laboratory test results during the screening phase:

   * Absolute neutrophil count ≤1.0 × 109 /L; (granulocyte colony stimulating factor use is permitted)
   * Hemoglobin level ≤7.5 g/dL (≤5 mmol/L); blood transfusions to maintain hemoglobin >7.5 are acceptable
   * Platelet count <75 × 109 /L for patients in whom <50% of bone marrow nucleated cells are plasma cells; otherwise platelet count <50 × 109 /L; no platelet transfusions in the past 7 days are allowed
   * Alanine aminotransferase (ALT) level ≥2.5 × upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) level ≥2.5 × ULN
   * Total bilirubin level ≥1.5 × ULN, (except for Gilbert Syndrome: direct bilirubin 2 × ULN)
   * Creatinine clearance ≤20 mL/min estimated using Cockcroft-Gault;
7. Has known allergies, hypersensitivity, or intolerance to monoclonal antibodies or human proteins, daratumumab or its excipients (refer to Investigator's Brochure), or known sensitivity to mammalian-derived products
8. Has plasma cell leukemia (>2.0 × 109 /L circulating plasma cells by standard differential), Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and/or skin changes), or amyloid light-chain amyloidosis
9. Is known or suspected of not being able to comply with the study protocol (e.g., because of alcoholism, drug dependency, or psychological disorder) or the patient has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient (e.g., compromise their well-being) or that could prevent, limit, or confound the protocol-specified assessments
10. Is considering becoming pregnant
11. Has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol- specified assessments
12. Has had major surgery within 2 weeks before C1D1, or will not have fully recovered from surgery, or has surgery planned during the time the patient is expected to participate in the study or within 2 weeks after the last dose of study drug administration. (Note: patients with planned surgical procedures to be conducted under local anesthesia may participate. Kyphoplasty is not considered a major surgery.)
13. Is eligible for stem cell transplant. Must be transplant ineligible as determined by their physician, or if transplant eligible, not expect to undergo transplant for at least 24 months after study enrollment.

NOTE: Investigators should ensure that all study enrollment criteria have been met at screening. If a patient's status changes (including laboratory results or receipt of additional medical records) after screening but before C1D1 such that he or she no longer meets all eligibility criteria, then the patient should be excluded from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CR) | 6 months
  percentage of patients who had complete response. Complete response is when patients achieve a negative immunofixation on the serum and urine and who also have an appearance of a soft tissue plasmacytomas and achieve less than or equal to 5 percent (%) plasma cells in the bone marrow.
Stringent Complete Response Rate (sCR) | 6 months
  percentage of patients who had stringent complete response. Patients with a stringent complete response in addition to the criteria that is required to have a complete response are required to have a normal free light chain ratio in the serum and absence of clonal cells in the bone marrow determined by either immunofluorescence or immunohistochemistry.
Safety of Selinexor plus DRd | 3 years
  frequency (incidence rate) of adverse effects

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 3 years
  percentage of patients who had either CR or sCR or very good partial response (VGPR) or partial response (PR).
Time to Next Treatment (TTNT) | 3 years
  the median interval between the date of study treatment initiation and the date of start of a new treatment
Duration of Response | 3 years
  the median time from first documented evidence of PR, CR,or sCR to date of progression or death or last date of contact for patients who did not progress or die
Progression-Free Survival (PFS) | 3 years
  the median time from randomization until the date of disease progression or death (by any cause in the absence of progression), regardless of whether the subject withdraws from the assigned study treatment
Overall Survival (OS) | 3 years
  the median time from randomization until death due to any cause or date of last contact for alive patients
Minimal Residual Disease (MRD) | 3 years
  number of patients who had CR or sCR and had: absence of phenotypically abnormal clonal plasma cells from bone marrow aspirates using Adaptive Technologies NGS Platform

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Rifkin, MD, FACP, Principal Investigator — US Oncology Research/McKesson Specialty Health
Locations (10):
- United States (10):
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - New York Oncology Hematology, P.C., Albany, New York
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Texas Oncology, P.A., Austin, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - Texas Oncology, P.A., San Antonio, Texas
  - Texas Oncology, P.A., Tyler, Texas
  - Virginia Cancer Specialists, PC, Gainesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data may be shared to other investigators in the form of publications, abstracts, and posters.